CLINICAL TRIAL: NCT00702988
Title: Pregnancy and Neonatal Follow-up of Ongoing Pregnancies Established During Clinical Trial 38826 for the Development of Org 36286 (Corifollitropin Alfa).
Brief Title: Pregnancy & Neonatal Follow-up of Ongoing Pregnancies Established During Clinical Trial 38826 (Study 38827)(P06056)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P06056; 38827
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy; Neonates
Keywords: Neonatal outcome; Congenital malformations; In-Vitro Fertilization; Controlled ovarian stimulation; Follow-up
MeSH Terms: conditions — Congenital Abnormalities | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group 1: all doses of Org 36286 (corifollitropin alfa) (60 μg, 120 μg and 180 μg)
  Interventions: Drug: Org 36286
- Experimental Group 2: 150 IU recFSH
  Interventions: Drug: recFSH

INTERVENTIONS:
Drug: Org 36286 — single dose of 60, 120, or 180 μg Org 36286 (experimental group administered under protocol 38826)
  Other Names: Corifollitropin alfa
  Groups: Experimental Group 1
Drug: recFSH — 150 IU recFSH daily (reference group administered under protocol 38826)
  Other Names: Follitropin Beta, Puregon®, Follistim®
  Groups: Experimental Group 2

SUMMARY:
The objective of this trial was to evaluate whether Org 36286 treatment for the induction of multifollicular growth in women undergoing controlled ovarian stimulation (COS) for in vitro fertilization (IVF) or intracytoplasmatic sperm injection (ICSI) is safe for pregnant subjects and their offspring.

DETAILED DESCRIPTION:
This was an open, prospective follow-up trial to monitor pregnancy, delivery, and neonatal outcome of women who became pregnant during Trial 38826. For this trial, no study specific assessments were required, but information obtained in standard practice was used.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who participated in Trial 38826 and became pregnant (as confirmed by USS at or beyond 10 weeks after ET) after having received at least one dose of either Org 36286 or Puregon®; and
* Able and willing to give written informed consent.

Exclusion Criteria:

* None

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with an ongoing pregnancy at least 10 weeks after embryo transfer in Trial 38826 were enrolled in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2003-10-01 (Actual); Primary Completion 2005-02-28 (Actual); Study Completion 2005-02-28 (Actual)

PRIMARY OUTCOMES:
Pregnancy status at 20 weeks of gestation | one pregnancy period
Take-home baby rate | one pregnancy period

SECONDARY OUTCOMES:
Pregnancy follow-up | one pregnancy period
Delivery follow-up | one pregnancy period
Neonatal outcome | one pregnancy period
Infant follow-up | one pregnancy period
Congenital malformations and chromosomal abnormalities | one pregnancy period

REFERENCES:
- [Derived] Bonduelle M, Mannaerts B, Leader A, Bergh C, Passier D, Devroey P. Prospective follow-up of 838 fetuses conceived after ovarian stimulation with corifollitropin alfa: comparative and overall neonatal outcome. Hum Reprod. 2012 Jul;27(7):2177-85. doi: 10.1093/humrep/des156. Epub 2012 May 15. PMID 22587997